CLINICAL TRIAL: NCT02029209
Title: To Predict Efficacy by Detecting Circulating Endothelial Cell Subsets and Blood Perfusion Parameters Changes in Vivo Tumor in the Phase II/III Study of Anlotinib in Patients With Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALTN-03-II 1.2-2
Record Dates: First submitted 2013-12-30; First posted 2014-01-07 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anlotinib (Experimental): Anlotinib QD orally and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Placebo Capsule (Placebo Comparator): Placebo capsule QD orally and it should be continued until disease progression or patients withdrawal of consent
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: Anlotinib — Anlotinib QD
  Arms: Anlotinib
Drug: Placebo Capsule — Placebo capsule QD
  Arms: Placebo Capsule

SUMMARY:
1. To reveal changes of peripheral markers and blood perfusion parameters in vivo tumor in the phase II study of anlotinib in patients with advanced non-small cell lung cancer.
2. To clarify the meaning of peripheral markers and blood perfusion parameters in vivo tumor in predicting the effect of anti-angiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology diagnosed with advanced NSCLC with measurable lesions;
2. Have failed for 2 lines of chemotherapy; 3.18-70 years,ECOG PS:0-2,life expectancy of more than 3 months;

4.Other cytotoxic drugs,radiation therapy,or surgery≥4 weeks; 5.Main organs function is normal; 6.Women of childbearing age should take contraceptive measures during the study and within 6 months after end.

Exclusion Criteria:

1. SCLC(including mixed with NSCLC);
2. The central cavity of Squamous cell carcinoma and hemoptysis with NSCLC;
3. Patients failed to use the anti-tumor angiogenesis therapy;
4. Patients have many influence factors toward oral medications ;
5. Brain metastases patients accompanied by symptoms or symptom control for less than two months;
6. Patients with severe and failed to controlled diseases,including: suboptimal blood pressure control;suffering from myocardial ischemia or above grade I myocardial infarction, arrhythmias and Class I heart failure;activity or failure to control severe infections;liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis;poorly controlled diabetes (FBG>10mmol/L);urine protein≥++,etc.
7. Patients failed to heal wounds or fractures for Long-term;
8. 4 weeks before enrollment, patients appeared NCI CTC AE grading >1 pulmonary hemorrhage; 4 weeks before enrollment, patients who appeared NCI CTC AE grade> 2 had other parts of the bleeding; patients have a tendency to bleed (e.g active peptic ulcer) or are receiving thrombolytic or anticoagulant therapy such as Warfarin, heparin or its analogues;
9. Patients occurred venous thromboembolic events within 6 months;
10. Patients who have HIV-positive or organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Number of circulating endothelial cell subsets（ total CECs 、 aCECs、apopCECs, etc.) | Different time points before and after treatment of anlotinib,an expected average of 3 weeks
  To detect number of circulating endothelial cell subsets（ total CECs 、aCECs、apopCECs, etc.) by Flow Cytometry;
The strength of intratumoral blood perfusion index (BV, BF, PS and MTT) . | Different time points before and after treatment of anlotinib,an expected average of 3 weeks
  To detect the strength of intratumoral blood perfusion index(BV, BF, PS and MTT) by CT perfusion imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Li Kai, doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- 20th Floor, Block C, Lake Road, Hexi District, Tianjin Medical University Cancer Institute and Hospital ., Tianjin, Tianjin Municipality, China